CLINICAL TRIAL: NCT00173732
Title: Establishment of Comprehensive Genetic Analysis From a Single Cell
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700629
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Preimplantation Genetic Diagnosis (PGD)
Keywords: Preimplantation genetic diagnosis (PGD); single cell; Multiple displacement amplification (MDA)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Preimplantation genetic diagnosis (PGD) is the integration of both assisted reproductive technologies and molecular genetic technologies and was shown to improve implantation rate and reduce spontaneous abortions after implantation. The principal problems in single cell PCR include amplification failure, ADO and contamination. Multiple displacement amplification (MDA) is a technique used in the amplification of very low amounts of DNA and reported to yield large quantities of high-quality DNA. By this approach, the diagnosis of gene disorders form single cell will be more accurate and reliable.

DETAILED DESCRIPTION:
Preimplantation genetic diagnosis (PGD) for couples at risk of conceptions with serious genetic disorders is firmly established as a valid reproductive option for couples to consider following appropriate genetic counseling. The procedure entails a balance of risks between establishing a successful pregnancy and minimizing the risk of misdiagnosis. PGD of single gene disorders relies on PCR-based tests performed on single cells (polar bodies or blastomeres). Despite the use of increasingly robust protocols, allele drop-out (ADO; the failure to amplify one of the two alleles in a heterozygous cell) remains a significant problem for diagnosis using single cell PCR. In extreme cases ADO can affect >40% of amplifications and has already caused several PGD misdiagnoses.

Fundamental to most genetic analysis is availability of genomic DNA of adequate quality and quantity. Because DNA yield from human samples is frequently limiting, much effort has been invested in developing methods for whole genome amplification (WGA) by random or degenerate oligonucleotide-primed PCR. However, existing WGA methods like degenerate oligonucleotideprimed PCR suffer from incomplete coverage and inadequate average DNA size. Multiple displacement amplification (MDA) provides a highly uniform representation across the genome. Amplification bias among eight chromosomal loci was less than 3-fold in contrast to 4-6 orders of magnitude for PCR-based WGA methods. Average product length was >10 kb. MDA is an isothermal, strand-displacing amplification yielding about 20-30 μg product from as few as 1-10 copies of human genomic DNA. Amplification can be carried out directly from biological samples including crude whole blood and tissue culture cells. MDA-amplified human DNA is useful for several common methods of genetic analysis, including genotyping of single nucleotide polymorphisms, chromosome painting, Southern blotting and restriction fragment length polymorphism analysis, subcloning, and DNA sequencing. MDA-based WGA is a simple and reliable method that could have significant implications for genetic studies, forensics, diagnostics, and long-term sample storage.

In this study we will carefully vary reaction conditions in single cell amplifications from isolated peripheral lymphocytes to minimize the rate of ADO. Consideration of the causal factors identified during this study should permit the design of PGD protocols that experience little ADO, thus improving the accuracy of PGD for single gene disorders.

ELIGIBILITY:
Inclusion Criteria:

* Preimplantation genetic diagnosis

Exclusion Criteria:

* nil

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Nan Lee, MD,PhD, Study Chair
Locations (1):
- Dept of Medical Genetics;National Taiwan University Hospital, Taipei, Taiwan